CLINICAL TRIAL: NCT00155064
Title: Kallikrein-kinin (KKS) and Renin-angiotensin-aldosterone System (RAAS) in Primary Aldosteronism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9361700632
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Hyperaldosteronism
Keywords: Primary aldosteronism; kallikrein; aldosterone; captopril
MeSH Terms: conditions — Hyperaldosteronism | interventions — Captopril; Losartan; Pharmaceutical Preparations

INTERVENTIONS:
Drug: captopril, Losartan (drug)

SUMMARY:
The tissue kallikrein-kinin (KKS) and renin-angiotension-aldosterone system (RAAS) had been implicated in regulating blood pressure and electrolyte homeostasis. Both of the KKS and RAAS may work coordinately to regulate salt metabolism, local blood flow. Thus, we conducted this study to elucidate, first, whether some alterations in components of the kallikrein-kinin system could do effect on aldosterone secretion.

Previous study has shown the post captopril plasma aldosterone concentration (PAC)/ plasma rennin activity (PRA) ration (ARR) was a reliable method for diagnosis of primary aldosteronism (PA). The ARR change by angiotensin II receptor blockade was reported to be significantly higher than that by ACE inhibitor. This study assessed whether angiotensin II receptor blockade offers any additional advantage in the diagnosis of PA. Clinically we evaluated the sensitivity and specificity of captopril (angiotensin-converting enzyme inhibition) and losartan (angiotensin II type 1 receptor blocker) test in PA patient. This interaction mechanism, in term, could further explain the interaction of KKS and RAAS.

DETAILED DESCRIPTION:
Hypertension affects 20% to 25% of adult population. Most patients are diagnosed as having essential or primary hypertension. Up to 10% to 15 % have an identifiable cause and many of those have an adrenal basis [Miroslava H. et al., 2002]. The tissue kallikrein-kinin (KKS) and renin-angiotension-aldosterone system (RAAS) had been implicated in regulating blood pressure and electrolyte homeostasis. Recent studies in humans indicate that the vasodilator tissue KKS, the counterpart of the tissue RAAS, is also expressed in the adrenal gland. The adrenal gland regulates sodium and water excretion and reabsorption through the release of aldosterone and corticosterone. Previous study reveals an anatomical linkage between the tissue KKS and sodium and water metabolism. Both of the KKS and RAAS may work coordinately to regulate salt metabolism, local blood flow. In contrast, although many investigators have supported the notion that Ang II and BK physiologically antagonize each other's effects on blood pressure, there are many instances where the two peptides exert common actions. For example, the Bradykinin also stimulates aldosterone release from adrenocortical cells through B2 receptors. Furthermore, the AT1 receptor and the bradykinin (B2) receptor form stable heterodimers, the two major signaling proteins triggered by AT1. In vitro studies (Margolius 1995) have shown that kallikrein acts as a prorenin-activating enzyme, and that tissue kallikrein can generate angiotensin II.

However, the interactions between both systems are complex and not always simply antagonistic. The interactions of the two systems on aldosterone secretion are not examined Thus, we conducted this study to elucidate, first, whether some alterations in components of the kallikrein-kinin system could do effect on aldosterone secretion.

Our study provides evidence that bradykinin contributes substantially to the aldosterone secretion with or without the effects of angiotensin. The data also could confirm whether ATR2-Bradykinin-B2-aldosterone really works. We want to realize the expression of angiotensin and bradykinin in the adrenal gland and hypertension related to these systems.

Previous study has showed the post captopril plasma aldosterone concentration (PAC)/ plasma rennin activity (PRA) ration (ARR) was a reliable method for diagnosis of primary aldosteronism (PA). The ARR change by angiotensin II receptor blockade was reported to be significantly higher than that by ACE inhibitor. This study assessed whether angiotensin II receptor blockade offers any additional advantage in the diagnosis of PA. Clinically we evaluated the sensitivity and specificity of captopril (angiotensin-converting enzyme inhibition) and losartan (angiotensin II type 1 receptor blocker) test in PA patient. This interaction mechanism, in term, could further explain the interaction of KKS and RAAS.

ELIGIBILITY:
Inclusion Criteria:

Patients with hypertension admitted for the diagnosis of primary aldosteronism

Exclusion Criteria:

Pregnant or lactating women. (Pre-menopause women, capable of bearing children will undergo pregnancy test), hypertension without discontinuous b-blocker, ACEI or ARB for more than 10 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of primary aldosteronism

SECONDARY OUTCOMES:
Subgroup analysis of primary aldosteronism

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, Md, PhD, Study Chair — National Taiwan University Hospital; Vin-Cent Wu, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Agharazii M, Douville P, Grose JH, Lebel M. Captopril suppression versus salt loading in confirming primary aldosteronism. Hypertension. 2001 Jun;37(6):1440-3. doi: 10.1161/01.hyp.37.6.1440. PMID 11408392
- [Background] Dendorfer A, Wolfrum S, Dominiak P. Pharmacology and cardiovascular implications of the kinin-kallikrein system. Jpn J Pharmacol. 1999 Apr;79(4):403-26. doi: 10.1254/jjp.79.403. PMID 10361880
- [Background] Hesse B, Rasmussen S, Lund JO, Christensen P, Damkjaer Nielsen M. Urinary excretion of kallikrein before and after operation for aldosterone-producing adenoma. Acta Med Scand. 1985;217(5):501-5. doi: 10.1111/j.0954-6820.1985.tb03253.x. PMID 3895826